CLINICAL TRIAL: NCT05864768
Title: Experimental Gingivitis in Omnivores and Vegetarians/Vegans. The Role of Diet in Periodontal Inflammation: A Controlled Clinical Study
Brief Title: The Role of Diet in Periodontal Inflammation: A Controlled Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Time Professor, G. d'Annunzio University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11012023
Record Dates: First submitted 2023-01-23; First posted 2023-05-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Periodontal Inflammation; Periodontal Diseases
Keywords: Experimental Gengivitis; Nutraceutical; Periodontal Inflammation
MeSH Terms: conditions — Periodontal Diseases | interventions — Diet, Vegan; Diet, Vegetarian

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a vegan/vegetarian diet (Experimental): After excluding patients with clinical signs of periodontitis, the patients recruited at baseline underwent prophylaxis and home oral hygiene instructions were given with brushing and flossing in order to reduce the parameters of inflammation and the presence of plaque (FMPS and FMBS). The use of antiseptics (chlorhexidine mouthwash 0.20%) was prescribed twice a day for 15 days.
  After 15 days from baseline (T0) all patients were recorded the parameters of FMPS, FMBS, PPD and Eastman Interdental Bleeding Index (EIBI) and were asked to stop using dental floss and mouthwash. All patients were recalled weekly 4 times after T0 (T1, T2, T3, T4) in order to monitor the parameters of inflammation and plaque accumulation by recording FMBS, FMPS and EIBI.
  Interventions: Dietary Supplement: Vegan/vegetarian diet
- Patients with an omnivorous diet (Active Comparator): After excluding patients with clinical signs of periodontitis, the patients recruited at baseline underwent prophylaxis and home oral hygiene instructions were given with brushing and flossing in order to reduce the parameters of inflammation and the presence of plaque (FMPS and FMBS). The use of antiseptics (chlorhexidine mouthwash 0.20%) was prescribed twice a day for 15 days.
  After 15 days from baseline (T0) all patients were recorded the parameters of FMPS, FMBS, PPD and Eastman Interdental Bleeding Index (EIBI) and were asked to stop using dental floss and mouthwash. All patients were recalled weekly 4 times after T0 (T1, T2, T3, T4) in order to monitor the parameters of inflammation and plaque accumulation by recording FMBS, FMPS and EIBI.
  Interventions: Dietary Supplement: Omnivorous diet

INTERVENTIONS:
Dietary Supplement: Vegan/vegetarian diet — At baseline, following the compilation of a periodontal chart in which pocket probing depth (PPD) and FMPS and FMBS were recorded, patients with pathological probing depths >3mm associated with periodontitis were excluded. Healthy patients underwent a prophylaxis session and oral hygiene instructions with brushing and flossing. A mouthwash based on chlorhexifdine 0.20% to be used twice a day was prescribed.
  At 15 days from the baseline (T0) the periodontal chart was compiled again and the parameters relating to PD, FMP, FMBS and the Eastman Interdental Bleeding Index (EIBI) were collected. Patients with FMBS and FMPS values >20% were excluded.
  From time T0 all patients were asked to suspend the interdental hygiene maneuvers by interrupting the use of dental floss and abandoning the use of mouthwash. All patients were recalled weekly, for a total of 4 times (T1, T2, T3, T4) in which parameters related to FMBS, FMPS and EIBI were recorded.
  Arms: Patients with a vegan/vegetarian diet
Dietary Supplement: Omnivorous diet — At baseline, following the compilation of a periodontal chart in which pocket probing depth (PPD) and FMPS and FMBS were recorded, patients with pathological probing depths >3mm associated with periodontitis were excluded. Healthy patients underwent a prophylaxis session and oral hygiene instructions with brushing and flossing. A mouthwash based on chlorhexifdine 0.20% to be used twice a day was prescribed.
  At 15 days from the baseline (T0) the periodontal chart was compiled again and the parameters relating to PD, FMP, FMBS and the Eastman Interdental Bleeding Index (EIBI) were collected. Patients with FMBS and FMPS values >20% were excluded.
  From time T0 all patients were asked to suspend the interdental hygiene maneuvers by interrupting the use of dental floss and abandoning the use of mouthwash. All patients were recalled weekly, for a total of 4 times (T1, T2, T3, T4) in which parameters related to FMBS, FMPS and EIBI were recorded.
  Arms: Patients with an omnivorous diet

SUMMARY:
Diet can influence the body's healing and repair mechanisms. A dietary imbalance obviously cannot trigger periodontal disease in the absence of a primum movens, which is bacterial plaque. However, it can condition its severity and extent by altering the permeability of the oral mucosa, the effectiveness of the immune response and the reparative potential of the gingival tissues.

Nutraceuticals is the science that studies the effects of the so-called food-drug, i.e. those foods that contain substances capable of performing a pharmacological function, modifying the functions of the organism. In particular, some molecules that are assimilated through various foods are able to penetrate the cell nucleus and influence, through an epigenetic mechanism, the expression or otherwise of some genes. The aim of our controlled study is to understand whether a vegetarian/vegan diet can be considered as protective for periodontal health compared to an omnivorous diet. For this purpose, we used a test group of 22 omnivorous subjects and a control group of 22 vegetarian/vegan patients in which experimental gingivitis was induced.

ELIGIBILITY:
Inclusion Criteria:

* Optimal systemic health conditions
* Non-Smoking
* Absence of cardio-vascular pathologies
* Absence of pulmonary pathologies
* Non-diabetic
* Not pregnant
* FMPS <20%
* FMBS <20%
* Omnivorous or vegan/vegetarian diet for at least a year
* Absence of periodontitis

Exclusion Criteria:

* Smokers
* Presence of systemic pathologies
* Presence of cardio-vascular disease
* Presence of periodontitis
* FMPS>20%
* FMBS>20%
* Pregnant women
* Presence of blood pathologies
* Taking medicines (hydantoins, nifedipine or cyclosporine)
* Taking oral contraceptives
* Bacterial, viral or fungal infections
* Idiopathic gingival fibromatosis
* Mucocutaneous disorders
* Allergic reactions to toothpastes and mouthwashes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Eastman Interdental Bleeding Index | Four weeks
  A wooden wedge is inserted buccally into the interdental space 2-3 mm, perpendicular to the long axis of the tooth, to assess for the presence of interdental inflammation (Yes/No).

SECONDARY OUTCOMES:
Pocket Probing Depth | Four weeks
  Change of the distance between the gingival margin and the depth of the probable site
Full Mouth Plaque Score | Four weeks
  Index that evaluates the general presence of bacterial plaque for all teeth. Through the passage of the probe, the presence of plaque deposits is reported for 4 surfaces for each tooth. A ratio is made between the contaminated surfaces and the total surfaces investigated to obtain a percentage value.
Full Mouth Bleeding Score | Four weeks
  Index that evaluates the general presence of bleeding for all teeth. Through the insertion of a periodontal probe, the presence of bleeding on probing is signaled for 4 sites for each tooth. A ratio is made between the bleeding sites and the total sites investigated to obtain a percentage value.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Paolantonio, MD; DDS, Principal Investigator — University G. D'Annunzio Chieti-Pescara
Locations (1):
- G. D'Annunzio University, Chieti, CH, Italy